CLINICAL TRIAL: NCT02230319
Title: Prevention of Paclitaxel Neuropathy With Cryotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Oncology & Hematology Associates of Northern Virginia (Other)
Collaborators: Inova Health Care Services (Other)
Responsible Party: Principal Investigator, Mary Wilkinson, Principle Investigator, Medical Oncology & Hematology Associates of Northern Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2014.1
Record Dates: First submitted 2014-08-25; First posted 2014-09-03 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: Cryotherapy; Cold therapy; Peripheral Neuropathy; Paclitaxel; Breast Cancer; Symptom management; Prevention
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases | interventions — Cryotherapy; Paclitaxel; Taxoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cryotherapy (Experimental): Each patient will receive cryotherapy administered during weekly paclitaxel treatments by Elasto gel™ Hypothermia mitts and slippers. Patients will wear the mitts and slippers for 15 minutes prior to treatment start, for 60 minutes during treatment, and for 15 minutes following treatment completion, for a total of 90 minutes.
  Interventions: Other: Cryotherapy; Drug: Paclitaxel

INTERVENTIONS:
Other: Cryotherapy
  Other Names: Cold therapy; Elasto gel™
Drug: Paclitaxel
  Other Names: Taxol; Taxanes

SUMMARY:
The purpose of this study is to determine if cryotherapy can effectively decrease the rate of neuropathy in patients undergoing weekly paclitaxel treatments.

ELIGIBILITY:
Inclusion Criteria

1. Women 18 years of age or older
2. Histologically or cytological proven diagnosis of breast cancer Stage I- III.
3. Must pl an to receive weekly paclitaxel treatment in either the adjuvant or neoadjuvant setting.
4. May have received prior treatment including, radiation, surgery chemotherapy hormone and biologics.
5. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
6. Patient signed informed consent.
7. Patient willing and able to comply with scheduled visits and treatment plan.

Exclusion Criteria

1. Patient presents with Grade 2 or greater peripheral neuropathy.
2. History of Raynaud's Disease.
3. Patient presents open or poorly-healing wounds on the hands or feet.
4. Patients with cold intolerance.
5. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment contraindicate patient participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 2 peripheral neuropathies induced by weekly paclitaxel. | From the date of randomization until date of first documented incidence of grade 2 peripheral neuropathy, assessed up to 2 years.

SECONDARY OUTCOMES:
Rate of completion of weekly adjuvant paclitaxel with the use of cryotherapy. | From the date of randomization until date of first documented incidence of grade 2 peripheral neuropathy, assessed up to 2 years.

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Wilkinson, MD, Principal Investigator — Medical Oncology & Hematology Associates of Northern Virginia
Locations (2):
- United States (2):
  - Medical Oncology & Hematology Associates of Northern Virginia, Fairfax, Virginia
  - Medical Oncology & Hematology Associates of Northern Virginia, Reston, Virginia